CLINICAL TRIAL: NCT06003439
Title: Virtual Reality for the Prevention and Cessation of Nicotine Vaping in Youth
Brief Title: Vaping Prevention and Vaping in Youth (Vapechat)
Acronym: Vapechat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-43102
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Vaping; Smoking Cessation
Keywords: Virtual reality (VR); High School Students
MeSH Terms: conditions — Vaping; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Health classes in each high school will be randomly assigned using a 1:3 threshold probability using a random digit generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Program (Experimental): Students in classrooms randomized to this group will receive the Virtual Reality vaping cessation and prevention program.
  Interventions: Behavioral: Virtual Reality Program; Behavioral: VR Program
- Assessment Only (No Intervention): Students in classrooms randomized to this group will not receive the VR intervention but will complete questionnaire assessment only.

INTERVENTIONS:
Behavioral: Virtual Reality Program — Behavioral: Virtual Reality Program The VR Program will be pre-installed on Meta Quest 2 headsets, which will be donned by students as a class to experience the intervention for approximately the length of one school class period (approximately 30-40 minutes). Each participant will experience the program once a week for 3 weeks. Participants who missed a week will complete the program by the 4th or 5th week.
  Other Names: VR Program
  Arms: Virtual Reality Program
Behavioral: VR Program — VR program participants will be able to download a mobile app that complements and reinforces the school-based VR session.
  Arms: Virtual Reality Program

SUMMARY:
Many youth are addicted to nicotine due to increased nicotine vaping (e.g., e-cigarettes). Unfortunately, there are no effective interventions to help teens quit vaping. In addition, existing vaping prevention programs have limited effectiveness because teens have reported that existing available interventions are out of touch with teen's culture and are not appealing to the intended audience. Therefore, to be effective, a vaping intervention must be acceptable, appealing, and engaging to teens, and most importantly, it should be designed to be channeled into an existing infrastructure such as the school setting.

The investigators' research group has designed a vaping prevention and cessation intervention that is implemented as a VR game for high school teens. The overall objective of this research is to assess the acceptability, feasibility, and preliminary efficacy of the VR experience among high school students in two high schools in Boston.

DETAILED DESCRIPTION:
The investigators will conduct a randomized trial of high school students (freshman to seniors) in the Boston area to determine feasibility, satisfaction, and preliminary efficacy of the VR-based vaping cessation and prevention game. Students will be randomized by class to either receive the Virtual Reality (VR) program (experimental condition) or control condition (questionnaire assessment only). There will be three VR sessions played at school during a health class. Participants in the VR condition will also engage in a gamified home-based component on their smartphone, in order to reinforce skills learned in the school-based VR experience.

Seven high school classes across two high schools will be randomized to VR intervention or assessment only. Health classes in each high school will be randomly assigned using a 1:3 threshold probability using a random digit generator. Participants will be enrolled in the study for approximately 6 weeks. In the first 3 weeks, participants will engage in the VR game experience once per week during their classes. In the fourth and fifth week, participants may make up any VR game session that they missed because of absence (e.g., illness). At week 6, participants will complete the follow-up questionnaire assessments.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled at Everett and Quincy High Schools (freshmen, sophomores, juniors, and seniors).
* Students in Health class
* Child assents

Exclusion Criteria:

* Teacher indicates that participation is not appropriate for the student (e.g., severe mental illness; visual or auditory disability; medical issue)
* Parent(s)/guardian(s) opt student out of the study.
* Prone to motion sickness or seizures.
* Visual impairments that would preclude playing VR or otherwise unable to use VR device.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Engagement with the VR program | 5 weeks
  Experimental condition arm. Playing time in minutes objectively measured by the program software; higher values mean a better outcome
Satisfaction with the VR game | 5 weeks
  Experimental condition arm. Self-report star rating of the VR game (1 to 5 stars); higher values mean a better outcome
Awareness of vaping | 5 weeks
  Experimental condition arm. Self-report awareness adapted from the Mobile App Rating Scale (MARS). Score range 1 - 5; higher values mean a better outcome
Knowledge of vaping | 5 weeks
  Experimental condition arm Self-report knowledge adapted from the Mobile App Rating Scale (MARS). Score range 1 - 5; higher values mean a better outcome
Attitudes towards vaping | 5 weeks
  Experimental condition arm. Self-report attitudes towards vaping adapted from the Mobile App Rating Scale (MARS). Score range 1 - 5; higher values mean a better outcome
Intention to change | 5 weeks
  Experimental condition arm. Self-report intention to change vaping behaviors adapted from the Mobile App Rating Scale (MARS). Score range 1 - 5; higher values mean a better outcome
Help seeking | 5 weeks
  Experimental condition arm. Self-report help seeking for vaping behaviors adapted from the Mobile App Rating Scale (MARS). Score range 1 - 5; higher values mean a better outcome
Gameplay experience and satisfaction | 5 weeks
  Experimental condition arm. Scores on a scale assessing the gameplay experience. Score range 1 - 4; higher values mean a better outcome

SECONDARY OUTCOMES:
Quit vaping attempts | 5 weeks
  Proportion of participants who have made one or more attempts to quit vaping for at least 24 hours
Past 30-days vaping frequency | 5 weeks
  Proportion of participants who have vaped '0', or '1-2', or '3-5', or '6-9', or '10-19', or '20-30' days in the past 30-days
Past 7-days vaping frequency | 5 weeks
  Proportion of participants who have vaped '0', or '1-2', or '3-4', or '5-6', or '7' days in the past 7-days
Frequency of current vaping | 5 weeks
  Proportion of participants who currently vape 'not at all', or 'some days', or 'most days', or 'every day'
Motivation to quit (or avoid) vaping within the next 30-days | 5 weeks
  Proportion of participants who are seriously thinking about quitting (or avoid) vaping within the next 30-days
Motivation to quit (or avoid) vaping | 5 weeks
  Scores on a scale assessing motivation to quit (or avoid) vaping. Score range 1 - 10; higher values mean a better outcome
Intention to try vaping (or quit vaping) | 5 weeks
  Proportion of participants who are 'probably not' or 'definitely not' thinking of vaping in the next 30- days
Confidence in avoiding vaping | 5 weeks
  Scores on a single item assessing confidence in avoiding vaping within 30-days. Scores range 1-10, higher values mean a better outcome
Self-efficacy to resist vaping | 5 weeks
  Scores on the adapted smoking abstinence self-efficacy questionnaire for adolescents. Scores range 0-24 , higher values mean a better outcome
Resilience | 5 weeks
  Scores on a brief resilience scale. Scores range 0-3 , higher values mean a worse outcome
Positive affect | 5 weeks
  Scores on the Pediatric Positive Affect (PROMIS) scale. Scores range 8-40, higher values mean a better outcome
Negative affect | 5 weeks
  Scores on the Negative Affect for Children scale Scores range 10-50, higher values mean a worse outcome
Tolerability of the VR game | 5 weeks
  Experimental condition arm Scores on the VR sickness questionnaire. Scores range 1-4, higher values mean a worse outcome
Intention to connect with vaping cessation resources | 5 weeks
  Scores on a single item assessing intentions to connect with vaping cessation resources. Scores range 1-10, higher values mean a better outcome
Emotion Regulation and Coping | 5 weeks
  Scores on the Adolescent-Coping Orientation for Problem Experience (A-COPE). Scores range 6-30, higher values mean a better outcome
Connection with vaping cessation resources | 5 weeks
  Proportion of participants who have made contact with any vaping cessation resources during the study

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Borrelli, PhD, Principal Investigator — Boston University, Goldman School of Dental Medicine, Center for Behavioral Science Research
Locations (1):
- Boston University, Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borrelli B, Weinstein D, Endrighi R, Ling N, Koval K, Quintiliani LM, Konieczny K. Virtual Reality for the Prevention and Cessation of Nicotine Vaping in Youths: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 15;14:e71961. doi: 10.2196/71961. PMID 40278000